CLINICAL TRIAL: NCT01961349
Title: A Multi-centre, Double-blind, Randomised, Parallel-group, Placebo-controlled, Phase III Confirmatory Study to Assess Efficacy and Safety of the Moderate Sedation of ICI35,868 With and Without EES0000645/A on Gastrointestinal Endoscopy
Brief Title: Phase III Study of ICI35,868 (Diprivan) With and Without EES0000645/A (SDS) on Gastrointestinal Endoscopy
Acronym: Kagami_SDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0092C00002
Record Dates: First submitted 2013-10-10; First posted 2013-10-11 (Estimated); Results first posted 2015-11-27 (Estimated); Last update posted 2015-11-27 (Estimated); Status verified 2015-10

CONDITIONS: Sedation to be Moderate for a Diagnostic Gastrointestinal Endoscopy and Gastrointestinal Endoscopic Polypectomy
Keywords: sedation, propofol, gastrointestinal endoscopy
MeSH Terms: interventions — soybean oil, phospholipid emulsion; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Placebo Comparator): Group 1 (placebo group) is treated by Anaesthesiologist
  Interventions: Drug: Intralipid
- Group 2 (Active Comparator): Group 2 (ICI35,868 without EES0000645/A) is treated by Anaesthesiologist
  Interventions: Drug: ICI35,868 (Diprivan)
- Group 3 (Active Comparator): Group 3 (ICI35,868 with EES0000645/A) is treated by Endoscopist
  Interventions: Drug: ICI35,868 (Diprivan) + EES0000645/A (SDS)

INTERVENTIONS:
Drug: Intralipid — Treated by Anaesthesiologist. (Intralipid is being used as a placebo for Diprivan.)
  Arms: Group 1
Drug: ICI35,868 (Diprivan) — Treated by Anaesthesiologist
  Arms: Group 2
Drug: ICI35,868 (Diprivan) + EES0000645/A (SDS) — Treated by Endoscopist with EES0000645/A(SDS)
  Arms: Group 3

SUMMARY:
This study is designed as a multi-centre, randomised, parallel-group, placebo-controlled, phase III confirmatory study. The study will be partially double-blinded: the comparison between Group 1 (placebo group) and Group 2 (ICI35,868 without EES0000645/A) will be carried out in double-blind, but the comparison between Group 1 (placebo group) and Group 3 (ICI35,868 with EES0000645/A) will be carried out in single-blind.

The efficacy and safety of ICI35,868 with and without EES0000645/A for the sedation to be moderate for a diagnostic gastrointestinal endoscopy and gastrointestinal endoscopic polypectomy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1.Provision of written informed consent prior to any study-related procedures/examinations 2.Aged 20 years and older 3.Subjects who are planned to undergo a non-emergent EGD or colonoscopy, including gastrointestinal endoscopic polypectomy that shall be completed within 1 hour (excluding the endoscopic submucosal dissection and ultrasonic endoscope, pernasal endoscope, etc.). Exclusion Criteria:

1. involvement in the planning and/or conduct of the study (applies to both sponsor's employees and/or staffs at the study site)
2. Subjects who underwent a endoscopic procedure under ICI35,868 (propofol) administration within 1 year.
3. Participation in another clinical study with an investigational product within 4 weeks prior to randomisation.
4. Baseline (Visit 1) of blood oxygen saturation (SpO2)<90% (room air)
5. ASA III, IV, V and VI ; Subject with serious disease of cardiovascular, respiratory, renal, liver, pancreatic or endocrine function.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Research Site, Moriya-shi
  - Research Site, Shinjuku-ku
  - Research Site, Yokohama

REFERENCES:
- See also: D0092C00002_CSR_Synopsis.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1892&filename=D0092C00002_CSR_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 279 consented subjects, 7 were excluded after screening.
Groups:
- Placebo: Placebo administered by the anaesthesiologist without EES0000645/A
- ICI35,868 Without EES0000645/A: ICI35,868 administered by the anaesthesiologist without EES0000645/A
- ICI35,868 With EES0000645/A: ICI35,868 administered and EES0000645/A operated by the GI physician or the nurse
Period: Overall Study
Arm/Group | Placebo | ICI35,868 Without EES0000645/A | ICI35,868 With EES0000645/A
Started | 54 | 107 | 111
Completed | 51 | 101 | 109
Not Completed | 3 | 6 | 2
Not completed — Withdrawal by Subject | 1 | 4 | 0
Not completed — Adverse Event | 0 | 0 | 1
Not completed — registration error, personal reason etc | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ICI35,868 Without EES0000645/A | ICI35,868 With EES0000645/A | Total
Number analyzed (Participants) | 51 | 101 | 109 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (14.3) | 55.4 (12.9) | 57.2 (14.8) | 56.8 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 36 | 34 | 87
  Male | 34 | 65 | 75 | 174

OUTCOME MEASURES:

1. Secondary Outcome: PSSI Total Score
Description: PSSI (Statistics of Patient Satisfaction with Sedation Instrument) total score obtained from 20 questions (1 to 7 points for each) adjusted to have range of 0 ( very dissatisfied: all items scored with 1 point) to 100 (very satisfied: all items scored with 7 points)
Time Frame: at 24-48 h after endoscopy
Population: FAS (Full Analysis Set)
Measure: Mean (Standard Deviation); unit: Score on a scale (0 - 100)
Arm/Group | Placebo | ICI35,868 Without EES0000645/A | ICI35,868 With EES0000645/A
Number analyzed (Participants) | 51 | 101 | 109
Score on a scale (0 - 100) | 65.3 (19.7) | 81.2 (12.5) | 80.8 (14.1)
Statistical Analysis 1: Comparison: Placebo vs ICI35,868 Without EES0000645/A; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Placebo vs ICI35,868 With EES0000645/A; Test type: Superiority or Other; p < 0.001, ANOVA

2. Primary Outcome: Achivement of Target Sedation
Description: The target sedation is defined as MOAA/S (Modified Observer's Assessment of Alertness/Sedation) scores 2 to 4 for ≥50% of all MOAA/S measurements from scope-in to scope-out.
Time Frame: from scope-in to scope-out
Population: FAS (Full Analysis Set)
Measure: Number (95% Confidence Interval); unit: % of patients
Arm/Group | Placebo | ICI35,868 Without EES0000645/A | ICI35,868 With EES0000645/A
Number analyzed (Participants) | 51 | 101 | 109
% of patients | 21.6 [11.3 to 35.3] | 88.1 [80.2 to 93.7] | 94.5 [88.4 to 98.0]
Statistical Analysis 1: Comparison: Placebo vs ICI35,868 Without EES0000645/A; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs ICI35,868 With EES0000645/A; Test type: Superiority or Other; p < 0.001, Fisher Exact

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | Placebo | ICI35,868 Without EES0000645/A | ICI35,868 With EES0000645/A
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/101 | 0/109
Other Adverse Events (participants affected / at risk) | 9/51 | 7/101 | 12/109
OTHER ADVERSE EVENTS (reported when occurring in more than 1.8% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=51) | ICI35,868 Without EES0000645/A (N=101) | ICI35,868 With EES0000645/A (N=109)
disinhibition (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
blood urine present (Investigations) | 1 (1) | 2 (2) | 3 (3)
sedation (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
oxygen saturation decreased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 5 (5) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less